CLINICAL TRIAL: NCT03150186
Title: Environmental Assessment of Secondhand Smoke Exposure in Private Settings and Outdoor Settings in Europe
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Public Health Agency of Barcelona (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); University of Aberdeen (Other); Istituto per lo Studio, la Prevenzione e la Rete Oncologica (Other); Universidad Politécnica de Cartagena (Other)
Responsible Party: Sponsor
Other Study IDs: TackSHS WP2
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Second Hand Tobacco Smoke
Keywords: second hand smoke; passive smoking; airborne nicotine; private settings; outdoors

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SHS exposure in homes: Measurement of nicotine level in private homes
  Interventions: Other: SHS exposure in homes
- SHS exposure in private cars: Measurement of nicotine level in private cars
  Interventions: Other: SHS exposure in private cars
- SHS exposure in outdoor settings: Measurement of nicotine level in outdoor settings (children playgrounds, terraces of hospitality venues, and entrances of primary school buildings)
  Interventions: Other: SHS exposure in outdoor settings

INTERVENTIONS:
Other: SHS exposure in homes — The investigators will recruit 20 non-smoking volunteers living in different homes with at least one smoker: 10 participants living in more deprived neighborhoods and 10 participants living in wealthier neighborhoods. Nicotine vapor phase will be measured using passive SHS samplers. The investigators will contact with participants and make an arrangement for measuring levels of nicotine at homes. First, the investigators will hang up a passive sampler in the main room of the house in accordance with the written protocol of sample collection. One week later, the investigators will come back to the house in a second visit to remove the sample. During the second visit the investigators will administer a specific questionnaire about environmental tobacco exposure to the participant.
  Groups: SHS exposure in homes
Other: SHS exposure in private cars — The investigators will measure levels of nicotine in 30 cars (two samples per car) in 2 European countries with different smoke-free legislation (Spain and UK). A convenience sampling will be performed considering feasibility. The investigators will recruit 30 drivers: 10 daily-smoking volunteers that usually smoke within their car; 10 daily-smoking volunteers that do not smoke within their car; and 10 non-smoking volunteers. To be eligible, participants have to spend a minimum of 30 minutes per day within the car. Nicotine vapor phase will be measured using passive SHS samplers. Two samplers will be hung up in each car during a period of 24 hours. One sampler will be open during the 24-hour sampling period. The other sampler will be only open during travelling time.
  Groups: SHS exposure in private cars
Other: SHS exposure in outdoor settings — In three types of outdoor settings (children playgrounds, terraces of hospitality venues, and entrances of primary school buildings), nicotine vapor phase will be measured using active SHS samplers. For each country, a convenience sampling of 60 outdoor settings (20 of each of the above mentioned settings) will be performed. Data collection will be conducted from March to October. The measurements will be able to be taken at any time of day providing that there are at least five adults. The investigators will collect nicotine samples using samplers attached to an air pump. Measurements will last 30 minutes. While measurements are being taken, data collectors will also conduct observations in accordance with the protocol of active sampling collection.
  Groups: SHS exposure in outdoor settings

SUMMARY:
This is a European study which is part of a larger research project (TackSHS project) funded by the European Union's Horizon 2020 Research and Innovation Programme (Grant Agreement 681040) and led by the Catalan Institute of Oncology. The main goal of the study is to assess the environmental levels of secondhand smoke (SHS) in non-regulated settings such as private and outdoor settings of 12 European countries (Bulgaria, France, Germany, Greece, Ireland, Italy, Latvia, Poland, Portugal, Romania, Spain and the United Kingdom) representing geographical, legislative (country-specific smoke-free policies) and cultural variations across Europe.

This is a multi-country cross-sectional study based on objective environmental measurements of SHS levels. Private settings studied are homes and cars and outdoors settings are terraces of hospitality venues, children playgrounds and entrances of primary school buildings. A total of 1,080 environmental measures of airborne nicotine will be collected. 20 environmental measures will be collected from homes and each of the outdoor settings for the 12 countries involved in the study (960 samples). Regarding cars, 60 environmental measurements will be collected in two countries (Spain and the UK) (120 samples), which have been selected taking into account differences in smoke-free legislation. Further information about SHS exposure will be collected for each setting through brief questionnaires or forms. Medians and interquartile ranges of nicotine concentrations will be calculated by country for each setting studied. Nicotine concentrations will be compared using non-parametric tests according to country, socioeconomic status and other determinants of exposure for each setting.

DETAILED DESCRIPTION:
OBJECTIVES

Main objective: to assess the levels of SHS in a range of private settings and outdoor settings in different European countries according to the type of setting, the smoke-free legislation and socioeconomic characteristics.

Specific objectives:

* To assess levels of SHS in homes and cars according to socioeconomic status
* To assess levels of SHS in outdoor settings (children playgrounds, terraces of hospitality venues and entrances of school buildings) according to socioeconomic status
* To analyze associations between air nicotine concentrations and self-reported information related to tobacco smoking and exposure to SHS in homes and cars
* To analyze associations between air nicotine concentrations and observational variables related to exposure to SHS in outdoor settings (children playgrounds, terraces of hospitality venues and entrances of school buildings)
* To assess relationships between levels of SHS and type of smoking legislation and socio-demographic characteristics across Europe according to different types of settings measured
* To develop evidence-based policy recommendations for policy makers and health authorities

METHODS

STUDY DESIGN

This is a multi-country cross-sectional study based on objective environmental measurements of SHS levels.

STUDY SETTINGS

The study will be carried out in private and outdoor settings in the following 12 European countries: Bulgaria, France, Germany, Greece, Ireland, Italy, Latvia, Poland, Portugal, Romania, Spain and the United Kingdom. Private settings studied will be homes and cars and outdoor settings will be terraces of hospitality venues, children playgrounds and entrances of primary school buildings.

SAMPLING

A total of 1,080 environmental measures will be collected. 20 environmental measures will be collected from homes and each of the outdoor settings for the 12 countries involved in the study (20 samples × 4 settings × 12countries = 960 samples). Regarding cars, 60 environmental measurements will be collected in two countries (Spain and UK) (120 samples), which have been selected taking into account differences in smoking legislation.

A convenience sampling will be performed considering feasibility and trying to include participants from different socioeconomic status (SES). Neighborhood SES will be measured using ecological synthetic SES indexes available in each country. Measures will be taken in private and outdoor settings located in the most deprived neighborhoods (those below the 20th percentile of the SES distribution) and the least deprived neighborhoods (those above the 80th percentile of the SES distribution).

FIELDWORK

Private settings: homes and cars

For each country, the investigators will measure levels of nicotine in 20 homes. We will recruit 20 non-smoking volunteers living in different homes with at least one smoker: 10 participants living in more deprived neighborhoods and 10 participants living in wealthier neighborhoods. Nicotine vapor phase will be measured during one week using passive SHS samplers. At the end of the week, the investigators will administer a specific questionnaire about SHS exposure to the participant.

The investigators will measure levels of nicotine in 30 cars (two samples per car) in two European countries with different smoke-free legislation (Spain and UK). A convenience sampling will be performed considering feasibility and trying to include participants with different smoking habits. The investigators will recruit 30 drivers: 10 daily-smoking volunteers that usually smoke within their car; 10 daily-smoking volunteers that do not smoke within their car; and 10 non-smoking volunteers. To be eligible, participants have to spend a minimum of 30 minutes per day within the car. Nicotine vapor phase will be measured using passive SHS samplers. Two samplers will be hung up in each car during a period of 24 hours. One sampler will be open during the 24-hour sampling period. The other sampler will be only open during travelling time. Outdoor settings: nicotine vapor phase will be measured using active SHS samplers. For each country, a convenience sampling of 60 outdoor settings (20 children playgrounds, 20 terraces of hospitality venues, and 20 entrances of primary school buildings) will be performed considering feasibility and trying to include the outdoor settings from different SES neighborhoods. Data collection will be conducted from March to October. The measurements will be able to be taken at any time of day providing that there are at least five adults. The investigators will collect nicotine samples using samplers attached to an air pump. Measurements will last 30 minutes. While measures are being taken, data collectors will also conduct observations in accordance with the protocol of active sampling collection. In each country, the investigators will measure levels of nicotine in 30 outdoor settings (10 playgrounds, 10 terraces of hospitality venues, and 10 entrances of primary school buildings) located in more deprived neighborhoods and 30 outdoor settings (as above) located in wealthier neighborhoods.

MAIN OUTCOMES

Vapour-phase nicotine (μg/m3) is the main objective outcome. The investigators will also register sample's code, location sampled, date and time when the monitor was installed and removed, time of tobacco exposure, volume of the area, smoke-free rules of the setting, and further relevant information related to the SHS exposure according to the different settings studied (e.g., for private settings: socio-demographic variables, intensity of tobacco exposure (number of smokers), minutes of exposure per day, number of cigarettes smoked per day, ventilation, use of air-conditioning or heating (only in cars), etc.; for outdoor settings: no smoking signs, presence of ashtrays and butts, smoke smell, number of people smoking, total number of adults and children, kind of venue, age group allowed to play (only in playgrounds), number of walls or roof (only in terraces), etc.).

DATA SOURCES

Environmental samples: Nicotine vapor phase will be measured using SHS samplers, which consist of a 37-mm diameter plastic cassette containing a filter treated with sodium bisulphate.

Passive samplers will be placed in private homes and cars. The samplers will be placed for a period of seven days in homes and of 24 hours in cars. In homes, samplers will be hung freely in the air approximately 2 meters high. They will not be placed where air does not circulate such as a corner, under a shelf or buried in curtains.

Active samplers will be used in outdoors settings. The samplers will be attached to an air pump with a flow rate ranging from 2 to 3 L/min, and 30-min measurements will be taken.

Questionnaire/Form: Questionnaires or forms will be fulfilled by trained personnel at the same time the samples are taken. There is a specific questionnaire or form to be filled for each setting. All questionnaires/forms gather some common questions and other specific questions according to the setting studied. Questionnaires/forms gather information on sampling area, date and time the samplers are placed and removed, the presence of tobacco smoking, specific characteristics of the setting studied, attitudes and behaviors towards tobacco, etc.

DATA MANAGEMENT

The study data will be kept in different databases according to the setting studied. Information obtained through forms and questionnaires will be entered on a computer by collaborators from each country. Then, all data bases will be encrypted and later on sent by e-mail to the ASPB. Individual forms and questionnaires will be scanned and sent electronically to the ASPB. Original versions will also be sent by post. All forms and questionnaires will be stored by the ASPB in agreement with the current law. Nicotine samples will be sent properly stored and identified to the ASPB during the fieldwork.

LAB ANALYSIS

All the nicotine samples will be analyzed by the laboratory of the Public Health Agency of Barcelona (Spain) using the gas chromatography/mass spectrometry method. Nicotine analysis will be conducted by the gas chromatography/mass spectrometry method, which has been officially accredited by the Spanish National Accreditation Entity (ENAC) according to ISO 17025 guidelines. This method allows quantifying the total amount of nicotine in the sample, with a lower limit of detection of 5 ng. Subsequently, the time weighted average nicotine concentration (μg/m3) can be estimated by dividing the amount of extracted nicotine by the volume of air sampled multiplied by the total number of minutes the filter has been exposed.

Blank samples will be analyzed for quality assurance and to assess potential contamination of the filters during manipulation of monitors, storage, shipment or shipment. A blank sample for each 20 samples will be analyzed.

STATISTICAL ANALYSIS

A first descriptive analysis will be conducted for all outcomes included in the study. Categorical variables will be described by raw frequencies and percentages and continuous variables will be described by means and standard deviations or medians and interquartile range (IQR). Medians and IQR of nicotine concentrations will be calculated by country for each setting studied. Box-plots will be used to visualize the distribution of nicotine concentrations. Nicotine concentrations obtained will be compared according to country, SES and other determinants of exposure for each setting, using non-parametric tests (the Mann Whitney U test or Kruskal-Wallis test as appropriate). Finally, correlations between nicotine concentration and variables related to the SHS recorded in the questionnaires or forms will be also assessed.

ETHICS

All participants taking part in environmental measurements collected in private settings (homes and cars) will be properly informed verbally and in writing, providing all pertinent information about the aims, methods, procedures, ethical issues and measures taken. Enrolling in the study will be voluntary and signing a written informed consent will be mandatory to take part in the study as agreement to participate. Informed consent will not be obtained to collect environmental measurements in outdoor settings. All written informed consents will be firstly stored in locked filing cabinets and principal investigators will be responsible for the informed consent of participants of their country. Later, written informed consent will be scanned, copied and sent electronically to the ASPB. All original informed consent will be post to the ASPB using a traceable mail courier. All original informed consent will be stored in accordance with Spanish legislation. All personal information will be treated as confidential and will be stored in agreement with the current laws. The study will be conducted in accordance with the Good Clinical Practice Guidelines of the Declaration of Helsinki and the current legal regulation about confidentiality of data.

INFORMED CONSENT

All informed consent will be written in English and in official language, according to the country involved in the project, to ensure potential participant's comprehension. The informed consent gathers information about the aims, methods and procedures of the study and properly informs about involvement of the participants and their rights as participants of the study. Two different specific informed consents have been designed according to the private setting (homes or cars) where the measurements are taken.

ELIGIBILITY:
Inclusion Criteria:

Homes:

* non-smoking volunteers living in different homes with at least one smoker
* participants living in more deprived neighborhoods (lower than 20th percentile of the SES distribution) or participants living in wealthier neighborhoods (above than 80th percentile of the SES distribution)

Cars:

* volunteers who travel in a car for at least 30min/day
* profiles of participants: 10 daily-smoking volunteers that usually smoke within their car; 10 daily-smoking volunteers that do not smoke within their car; and 10 non-smoking volunteers.

Outdoor settings:

* there should be at least five adults present at the moment of the measurement start
* the settings should be located in more deprived neighborhoods (lower than 20th percentile of the SES distribution) or in wealthier neighborhoods (above than 80th percentile of the SES distribution)
* playgrounds with slides, swings or other similar playing equipment and located outdoors (for children playgrounds)
* terraces with at least one wall or roof, placed in cafeterias, bars or night pubs (for terraces)

Exclusion Criteria:

* volunteers with literacy level or language skills preventing them from understanding the study documents

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Private homes, private cars, three types of outdoor settings (terraces of hospitality venues (1), children playgrounds (2) and entrances of primary school buildings (3) in 12 European countries
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
SHS exposure in private and outdoor settings | Passive sampling (homes and cars): 1 week in homes and 24 hours in cars; active sampling (outdoor settings): 30 minutes
  Vapour-phase nicotine (μg/m3) measured via passive sampling in private homes and cars and via active sampling in three types of outdoor settings.

CONTACTS AND LOCATIONS:
Overall Officials: Maria J López, PhD, Principal Investigator — Public Health Agency of Barcelona
Locations (1):
- Agència de Salut Pública de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: TackSHS Project — http://tackshs.eu/